CLINICAL TRIAL: NCT03455400
Title: Ventilation Distribution Observed With Electrical Impedance Tomography (EIT) During Spontaneous Breathing in Healthy Newborn Infants
Brief Title: Ventilation Distribution During Spontaneous Breathing in Healthy Newborn Infants
Status: Completed | Type: Observational
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Other Study IDs: EETTMK:104/2017
Record Dates: First submitted 2018-02-27; First posted 2018-03-06 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Spontaneous Breathing; Full-Term Neonate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Swisstom BB2 EIT device — Swisstom BB2 EIT device with NEO SensorBelts will be used to measure ventilation distribution during spontaneous breathing and position changes in healthy newborn infants.

SUMMARY:
Electrical impedance tomography (EIT) is an evolving monitoring tool for respiratory support in neonatal and pediatric intensive care. In this observational study basic EIT parameters will be measured on 20 healthy newborn infants during spontaneous breathing and assess the effect of position changes in ventilation distribution.

DETAILED DESCRIPTION:
NEO SensorBelts will be used to observe ventilation distribution in healthy newborn infants during quiet spontaneous breathing. Child's position will be changed 5 times every 10 minutes in a random order. Positions observed will be: left lateral, right lateral, supine, prone face to left, prone face to right and supine with the bed tilted 30 degrees. Total duration for the recording will be 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from a parent or legal guardian
* Gestational age 37+0 - 42+0 weeks
* Uneventful follow-up in maternity ward

Exclusion Criteria:

* Respiratory distress
* Admission to NICU
* Thorax skin lesions
* Prior participation in this study

Ages: 12 Hours to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 20 healthy full-term infants
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Anteroposterior ventilation distribution | 1 hour
  The ventral-to-dorsal center of ventilation will be calculated as described in (Frerichs et al., Acta AnaesthesiolScand. 1998; 42:721-726) as a value between 0 and 100%, higher values indicating a more dorsal distribution of ventilation.
Right-to-left ventilation distribution | 1 hour
  Changes in right-to-left ventilation distribution following position changes will be calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No